CLINICAL TRIAL: NCT03541291
Title: Utility of MRI With Doppler Ultrasound Gating for Advanced Fetal Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mike Seed, Qualified Investigator, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1000055684
Record Dates: First submitted 2018-05-18; First posted 2018-05-30 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMART-SYNC LM03 (Experimental): All participants
  Interventions: Device: SMART-SYNC LM03

INTERVENTIONS:
Device: SMART-SYNC LM03 — Doppler ultrasound cardiac gating device for fetal MRI application

SUMMARY:
We will test an ultrasound device that uses sound waves to detect the fetal heart beat, and use this device to tell the MRI scanner when to collect pictures of the fetal heart. This will help freeze motion of the fetal heart, to make MRI pictures sharper. This will be important for assessing human fetal heart disease, an active area of research at our institution.

ELIGIBILITY:
Inclusion Criteria:

* pregnant adults (age 18 and up) with fetus affected by congenital heart disease
* singleton pregnancy in their 2nd and 3rd trimesters
* scheduled for a clinical fetal ultrasound examination at the Fetal Echocardiography Clinic at SickKids

Exclusion Criteria:

* claustrophobia
* cardiac pacemaker
* non-MRI compatible implants
* non-singleton pregnancy
* obesity (BMI > 30)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Comparison between fetal MRI and fetal echocardiography | within 2 weeks of participation in the study
  Anatomic MR images of the fetal heart will be acquired using prospective gating information from the Doppler ultrasound probe (SMART-SYNC LM03) and used to calculate ejection fraction. These values will be compared with corresponding reference values obtained during the patient's visit to the Fetal Echocardiography Clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seed, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-09-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03541291/Prot_001.pdf